CLINICAL TRIAL: NCT03454191
Title: Efficacy of Erector Spinae Plane Block for Postoperative Analgesia in Adult Patients Undergoing Thoracoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment stopped due to lack of research assistant
Sponsor: Eric Albrecht (Other)
Responsible Party: Sponsor-Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2017-01772
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (Experimental)
  Interventions: Procedure: Erector spinae plane block
- Placebo (Placebo Comparator)
  Interventions: Procedure: No injection

INTERVENTIONS:
Procedure: Erector spinae plane block — Injection of local anaesthetics below the erector spinae muscle after induction of anaesthesia
  Arms: Erector spinae plane block
Procedure: No injection — No injection
  Arms: Placebo

SUMMARY:
The erector spinae plane block has been recently described as an effective analgesic postoperative pain treatment in case reports. It consists of injecting local anaesthetics below the erector spinae muscle, at the level of the transverse processes, in order to anaesthetize the thoracic roots coming out from the spinal cord. However, the analgesic efficacy has never been demonstrated in a randomized controlled trial. Therefore, the objective of this study is to investigate the analgesic benefit of this block on patients scheduled for thoracoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoscopy
* physical status I-III

Exclusion Criteria:

* allergy to local anaesthetics
* other contraindications to peripheral nerve blocks
* patients suffering from chronic pain condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
IV morphine consumption | 24 postoperative hours
  mg

SECONDARY OUTCOMES:
IV morphine consumption | 2 postoperative hours
  mg
IV morphine consumption | 48 postoperative hours
  mg
Pain scores | 2, 24, 24 postoperative hours
  Visual analog scale, 0-10
Chronic pain scores | 3 and 6 postoperative months
  Visual analog scale, 0-10
Forced vital capacity | 24 and 48 postoperative hours
  L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Centre Hospitalier Universitaire Vaudois and University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR